CLINICAL TRIAL: NCT04687787
Title: Comparison of Core Stabilization Exercises and Routine Exercise Therapy on Pregnancy Induced Pelvic Girdle Pain
Brief Title: Core Stabilization Versus Routine Routine Exercises in Pelvic Girdle Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec/00837 Zahra Ejaz
Record Dates: First submitted 2020-12-25; First posted 2020-12-29 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Pelvic Girdle Pain
Keywords: Core Stability Exercises; Pelvic Girdle Pain; Pregnancy; Physical therapy management
MeSH Terms: conditions — Pelvic Girdle Pain

STUDY DESIGN:
Intervention Model Description: There will be two groups which will receive physical therapy interventions. one will be experimental and other will be control group.
Who Masked: Participant
Masking Description: Participants will be kept blind of the treatment provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): This group will receive Core Stability Exercises with Application of TENS
  Interventions: Other: Core Stabilization exercises
- Group II (Active Comparator): This group will receive Routinely prescribed Exercises with application of TENS
  Interventions: Other: Routinely prescribed exercises

INTERVENTIONS:
Other: Core Stabilization exercises — . Each session will be given for 40 mins (20 mins for TENS and 20 Mins for exercise) Core Stability Exercises include Kegel Exercises, Modified V-sit, opposite Arm Leg Raise, Seated Side bends poses, Dumbell Side bends and Pelvic Tilt. Participants will perform 1 set of exercise having 10 repetitions with hold of 5 seconds. Session would be performed thrice a week.
  Arms: Group I
Other: Routinely prescribed exercises — Each session will be given for 40 mins ( 20 mins for TENS and 20 Mins for exercise Routinely prescribed exercises composed of Hamstring stretches, hip flexor stretches, hip extensor stretches, calf stretches, and back extensor stretches. Participants will perform 1 set of exercise having 10 repetitions with hold of 5 seconds. Session would be performed thrice a week.
  Arms: Group II

SUMMARY:
Pregnancy Induced Pelvic Girdle Pain (PGP) is common complaint in pregnant women all over the world and it has a major impact on health and functioning as it decreases quality of life. The onset of PGP is usually seen at 17-19 week of gestation, with a peak of incidence at 24- 36 weeks. The purpose of this study is to compare the effects of stabilization exercises on pregnancy induced pelvic girdle pain and its effects on the activity levels as compare to the physiotherapy exercises that are routinely prescribed

DETAILED DESCRIPTION:
the study is Randomized Controlled trial which will be conducted in the Outpatient Physical therapy Department. Patient with suspected PGP will be referred by midwives, physicians or directly contact to Physiotherapist. Sample size of 30 individual was calculated by using open Epi tool with 95% confidence Interval (CI) and 80% Power. Inclusion criteria for patients is 13-28 gestational weeks determined by special test include P4 Test (Posterior Pelvic Pain Provocation) and FABER test (Flexion Abduction and External Rotation). Individuals would be randomly allocated into two groups by sealed envelope method.

Assessment will be done at base line and 4th week by using NPRS and PGP Questionnaire. Data will be analyzed by using SPSS version 21.

ELIGIBILITY:
Inclusion Criteria:

* Women having Pelvic Girdle Pain in 2nd trimester or 1st month of third trimester.
* Age between 20-40 years.
* Positive FABER test (leg of patient is placed in figure of 4 and apply small amplitude oscillation are applied at end range of motion after stabilizing opposite side of Pelvis.

Positive test elicits pain and limited ROM)

* Positive P4 test (leg of patient is flexed at 90 degrees in supine position. Sacrum is stabilized by one hand and axial pressure is applied along the femur by other hand.

Positive test elicits pain in SI joint).

Exclusion Criteria:

* History of Pelvic Fractures and Surgery
* History of metabolic diseases.
* Radiculopathy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only pregnant females will be recruited in the study
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | Baseline
  Numeric pain rating scale (NPRS) is an 11 point (0-10) Scale used to measure pain. Patient verbally select value between (0-10) on the basis of intensity of pain. (0) means No pain and (10) means maximum pain experienced at baseline.
Numeric pain rating scale (NPRS) | Post 4 week
  Numeric pain rating scale (NPRS) is an 11 point (0-10) Scale used to measure pain. Patient verbally select value between (0-10) on the basis of intensity of pain. (0) means No pain and (10) means maximum pain experienced at baseline.
Pelvic Girdle Pain Questionnaire (PGPQ) | Baseline
  The Pelvic Girdle Questionnaire (PG Q) is a condition-specific measure for women with pelvic girdle pain (PGP). The questionnaire has 25 items under two sub-scales (20 items for activates and 5 items for symptoms), with percentage scores that range from 0 (no disability) to 100 (great disability).
Pelvic Girdle Pain Questionnaire (PGPQ) | Post 4 weeks
  The Pelvic Girdle Questionnaire (PG Q) is a condition-specific measure for women with pelvic girdle pain (PGP). The questionnaire has 25 items under two sub-scales (20 items for activates and 5 items for symptoms), with percentage scores that range from 0 (no disability) to 100 (great disability).

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Alam Family Hospital, Rawalpindi, Punjab Province
  - Izzat Ali Shah Hospital, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almousa S, Lamprianidou E, Kitsoulis G. The effectiveness of stabilising exercises in pelvic girdle pain during pregnancy and after delivery: A systematic review. Physiother Res Int. 2018 Jan;23(1). doi: 10.1002/pri.1699. Epub 2017 Nov 8. PMID 29115735
- [Background] Walters C, West S, A Nippita T. Pelvic girdle pain in pregnancy. Aust J Gen Pract. 2018 Jul;47(7):439-443. doi: 10.31128/AJGP-01-18-4467. PMID 30114872
- [Background] Timothy J. Piper EJ, Mike Haiduke, Mike Waller, and Cathy McMillan. Core Training Exercise Selection During Pregnancy. Strength and Condtioning Journal. 2012;34(1).
- [Background] Saleh MSM, Botla AMM, Elbehary NAM. Effect of core stability exercises on postpartum lumbopelvic pain: A randomized controlled trial. J Back Musculoskelet Rehabil. 2019;32(2):205-213. doi: 10.3233/BMR-181259. PMID 30282349
- [Background] Akhtar MW, Karimi H, Gilani SA. Effectiveness of core stabilization exercises and routine exercise therapy in management of pain in chronic non-specific low back pain: A randomized controlled clinical trial. Pak J Med Sci. 2017 Jul-Aug;33(4):1002-1006. doi: 10.12669/pjms.334.12664. PMID 29067082